CLINICAL TRIAL: NCT01445990
Title: Evaluation of Free Tissue Flaps Viability With Capillary Glucose and Lactate Measurements Compared With Clinical Examination
Brief Title: Efficacy Study of Free Flap Monitoring Using Capillary Lactate and Glucose Measurements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Narcisse Zwetyenga (Other)
Collaborators: Centre Hospitalier Universitaire de Besancon (Other); Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor-Investigator, Narcisse Zwetyenga, Head of Maxillo-Facial, Plastic and Reconstructive Surgery Unit, Centre Hospitalier Universitaire Dijon
Organization: Centre Hospitalier Universitaire Dijon (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2009-A01262-55
Record Dates: First submitted 2011-09-30; First posted 2011-10-04 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-10

CONDITIONS: Postoperative Complications
Keywords: free tissue flaps; lactic acid; glucose; thrombosis; diagnostic test; Pedicle postoperative complications diagnosis
MeSH Terms: conditions — Postoperative Complications; Thrombosis

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Lactate-meter: LactatePro (ARKRAY Inc) — Capillary glucose and lactate measurement. Every hours for the first 24 hours, and every 4 hours for the next 4 days.

SUMMARY:
Evaluation of capillary glycaemia and lactataemia measurements for pedicle impairments diagnosis in free tissue transfers is realized.

These measures are done after surgical reconstructions with free tissue flap, simultaneously with clinical examination. These biological data aren't available to make clinical diagnosis of complication; only clinical examination is allowed in this way.

A posteriori, clinical and biological parameters will be compared in order to determine if capillary glycaemia and lactataemia measurements is a good procedure for free tissue flaps monitoring.

DETAILED DESCRIPTION:
Free tissue flap reconstruction has become a reliable technique. Nevertheless, pedicle thrombosis is dreaded, and the earlier the diagnosis of such complications is made, the higher the surgical salvage rate is.

Clinical monitoring remains the most useful and used monitoring method, but makes late and unreliable diagnosis. Numerous studies are searching for ideal monitoring technics with regard to free flaps. Nowadays, the most efficient ones often deal with expensive and invasive technics. In this study, capillary lactataemia and glycaemia measurements are evaluated for pedicle impairments diagnosis.

Measurements of these 2 biological parameters seem to be a powerful screening test of pedicle impairments in microdialysis. But these parameters are measured in this case in interstitial tissues. Capillary measurements will probably provide different results, and needs to be evaluated.

For that purpose, surgical reconstructions with free tissue flap will be clinically monitored during five days, every hours for the first 24 hours, and every 4 hours for the next 4 days. Simultaneously, blind measurements of capillary lactataemia and glycaemia will be performed. Biological and clinical data will be systematically written in the corresponding table of the individual register together with the time the examination is done.

In this register, all complications and evolutions of the flaps will be recorded.

A posteriori, parallel between clinical and biological events will be studied. This multicenter prospective study will show first if capillary measurements of glucose and lactate permit to screen pedicle complications of free flaps. In case of efficacy of this technique, thresholds of glucose and lactate permitting such diagnoses will be calculated in order to define a sensitive screening test. Moreover, temporal differences between clinical and biological diagnoses of pedicle impairments will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Informed patient
* Signed informed consent
* Free tissue flap reconstruction
* Accessible flap for measurements

Exclusion Criteria:

* Pregnancy
* Patient under 18
* Unaccessible flap

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Clinical examination of the flap | Beginning immediately after free flap surgical procedure. Realized 48 times during the 5 first postoperative days. Synchronous with capillary glucose and lactate measurements.
  Clinical examination is done immediately after the end of the surgical procedure (Expected 1 to 5 hours after the end of arterial anastomosis).
  Then, examinations are done every hours for the first 24 hours, and every 4 hours for the next 4 days.
  The clinical examination was standardized: skin paddle colour and temperature, skin reperfusion time, and bleeding test with a prick.
  In order to avoid bias, examinations are performed by caregivers before capillary lactate and glucose measurements, and they hadn't any information about expected results of lactate and glucose values.

SECONDARY OUTCOMES:
Capillary lactate measurements | Beginning immediately after free flap surgical procedure. Realized 48 times during the 5 first postoperative days. Synchronous with capillary glucose measurements and clinical examinations.
  Capillary lactate is measured immediately after the end of the surgical procedure (Expected 1 to 5 hours after the end of arterial anastomosis).
  Then, measurements are done every hours for the first 24 hours, and every 4 hours for the next 4 days.
  In order to avoid bias, measurements are performed by caregivers after clinical examination, and they hadn't any information about expected results of lactate and glucose values.
Capillary glucose measurements | Beginning immediately after free flap surgical procedure. Realized 48 times during the 5 first postoperative days. Synchronous with capillary lactate measurements and clinical examinations.
  Capillary glucose is measured immediately after the end of the surgical procedure (Expected 1 to 5 hours after the end of arterial anastomosis).
  Then, measurements are done every hours for the first 24 hours, and every 4 hours for the next 4 days.
  In order to avoid bias, measurements are performed by caregivers after clinical examination, and they hadn't any information about expected results of lactate and glucose values.

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Henault, MD, Study Chair — Centre Hospitalier Universitaire Dijon; Narcisse Zwetyenga, PhD, Principal Investigator — Centre Hospitalier Universitaire Dijon; Julien Pauchot, MD, Study Chair — Centre Hospitalier Universitaire Dijon; Raphaël Sinna, MD, Study Chair — Centre Hospitalier Universitaire, Amiens; Christophe Meyer, PhD, Study Chair — Centre Hospitalier Universitaire, Besançon
Locations (4):
- France (4):
  - Department of Plastic reconstructive and Aesthetic Surgery. University Hospital Amiens, Amiens
  - Maxillo-Facial Surgery, Besancon Univestitary Hospital, Besançon
  - Orthopaedic, Traumatologic and Plastic Surgery Unit, Besancon Universitary Hospital, Besançon
  - Maxillo-Facial, Plastic and Reconstructive Surgery Unit, Centre Hospitalier Universitaire, Dijon